CLINICAL TRIAL: NCT01298232
Title: One-year Outcomes of Electromechanical Activation Time (EMAT)-Guided vs. Symptom-guided Heart Failure Therapy in Acute Heart Failure Syndrome (AHFS) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Taipei Veterans General Hospital, Taipei Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 100-01-001C
Record Dates: First submitted 2011-02-15; First posted 2011-02-17 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMAT-guided therapy (No Intervention): electromechanical activation time (EMAT, obtain by phonocardiogram, Audicor, USA)
  Interventions: Other: Cardiophonogram
- Symptomatic-guided therapy (No Intervention): HF therapy guided by clinical symptoms
  Interventions: Other: Cardiophonogram

INTERVENTIONS:
Other: Cardiophonogram — Using data from cardiophonogram, the EMAT and S3 intensity, to guided clinical therapy for acute heart failure

SUMMARY:
Left ventricular systolic time intervals, including pre-ejection period (PEP), ejection time (ET), and their ratio (PEP/ET), is determined by the systolic and diastolic function and ventriculo-arterial coupling. The investigators have shown the usefulness of the electromechanical activation time (EMAT, equals PEP minus isovolumic contraction time) in the prediction of cardiac mortality or re-hospitalization for heart failure in patients with the acute heart failure syndrome (AHFS). Therefore, the objective of the present proposal is to compare 12-month outcomes of EMAT-guided vs symptom-guided heart failure therapy in patients with AHFS.

DETAILED DESCRIPTION:
Left ventricular systolic time intervals, including pre-ejection period (PEP), ejection time (ET), and their ratio (PEP/ET), is determined by the systolic and diastolic function and ventriculo-arterial coupling. The investigators have shown the usefulness of the electromechanical activation time (EMAT, equals PEP minus isovolumic contraction time) in the prediction of cardiac mortality or re-hospitalization for heart failure in patients with the acute heart failure syndrome (AHFS). Therefore, the objective of the present proposal is to compare 12-month outcomes of EMAT-guided vs symptom-guided heart failure therapy in patients with AHFS.

A total of 120 patients aged 18 years or older and hospitalized at Taipei Veterans General Hospital or National Taiwan University Hospital due to AHFS will be enrolled in three years, and randomized into 2 treatment strategies, that is, intensified (EMAT-guided) therapy or standard (symptom-guided) therapy. Systolic time intervals and EMAT normalized by cardiac cycle length (%) are measured separately by separate automated acoustic devices. All parameters will be assessed within 24 hours before discharge, and at 2 weeks, and 3, 6, and 12 months after discharge. Patients randomized to the EMAT-guided group will undergo intensified therapy of heart failure with the goal to reduce both %EMAT<15 and symptoms to NYHA ≤II. Patients randomized to the symptom-guided group will have standard medical care, with the goal to reduce symptoms to NYHA ≤II. The primary efficacy variable is defined as the time to cardiovascular death or heart failure hospitalization within 1 year after randomization. This study will be the first prospective randomized controlled trial to study the management of patients with AHFS using EMAT and will provide unique information comparing two treatment strategies irrespective of natriuretic peptides regarding prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are hospitalized due to AHFS and have a plasma NT-proBNP ≥ 1600 pg/ml at admission.
2. Patients give written consents to participate in the study.

Exclusion Criteria:

1. Patients with an implanted pacemaker.
2. Patients with chronic kidney disease, stage 5 and warranted dialysis.
3. Patients with hypertrophic obstructive cardiomyopathy.
4. Patients with cardiac temponade or constrictive pericarditis.
5. Acute coronary syndrome, stroke, transient ischemic attack, cardiac, carotid or major vascular surgery, percutaneous coronary intervention (PCI) or carotid angioplasty, within the past 1 months prior to index hospitalization.
6. Coronary or carotid artery disease likely to require surgical or percutaneous intervention within the 6 months after discharge at index hospitalization.
7. Patients with left ventricular assistance device (LVAD device).
8. Documented ventricular arrhythmia with syncope episodes within past 3 months, prior to index hospitalization that is untreated.
9. Symptomatic bradycardia or second or third degree heart block without a pacemaker.
10. Implantation of a CRT (cardiac resynchronization therapy) device within the prior 1 month before index hospitalization or intent to implant a CRT device.
11. Presence of hemodynamically significant mitral and/or aortic valve disease, except mitral regurgitation secondary to left ventricular dilatation.
12. Presence of other hemodynamically significant obstructive lesions of left ventricular outflow tract, including aortic and sub-aortic stenosis.
13. Severe primary pulmonary, renal or hepatic disease.
14. Presence of any other disease with a life expectancy of < 1 year.
15. Subjects get pregnant or will be pregnant within 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular mortality and heart failure rehospitalization | within 1 year after discharge

SECONDARY OUTCOMES:
All-cause mortality | within 1 year after discharge

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - National Taiwan University Hsopital, Taipei
  - Taipei Veterans General Hospital, Taipei

REFERENCES:
- [Derived] Sung SH, Huang CJ, Cheng HM, Huang WM, Yu WC, Chen CH. Effect of Acoustic Cardiography-guided Management on 1-year Outcomes in Patients With Acute Heart Failure. J Card Fail. 2020 Feb;26(2):142-150. doi: 10.1016/j.cardfail.2019.09.012. Epub 2019 Sep 27. PMID 31568829